CLINICAL TRIAL: NCT05314114
Title: Selective Omission of Axillary Surgery in Distinct Responders With Triple-negative and HER2-positive Breast Cancer After NACT
Brief Title: Selective Omission of Axillary Surgery in Triple-negative and HER2-positive Breast Cancer After NACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Professor, Director of the Breast Cancer Department, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-P29
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No Axillary Surgery (Experimental): No axillary surgery including SLNB
  Interventions: Procedure: No axillary surgery

INTERVENTIONS:
Procedure: No axillary surgery — No axillary surgery

SUMMARY:
Neoadjuvant chemotherapy (NACT) is standard treatment for many triple-negative (TNBC) and HER2-positive breast cancer. Study showed about half of the biopsy-proven axillary disease will be eradicated by NACT and converted to ypN0 indicating the efficacy of systemic treatment in local disease control.

According to current guidelines, all initial cN0 patients will undergo sentinel lymph node biopsy (SLNB) after NACT and further axillary dissection (ALND) if tumor residual is discovered after SLNB. Data suggest patients who underwent SLNB have a significantly higher rate of disability in the early post-operative period compared to patients who did not and the avoidance of SLNB might translate into a considerable reduction of physical and emotional distress. Recent studies revealed the association between breast pCR and ypN0 status after NACT. Initially cN0 TNBC and HER2-positive breast cancer patients who achieve pCR in breast after NACT have a very low risk of positive lymph node residual and are very unlikely to benefit from further axillary surgery including SLNB.

The investigators designed a clinical trial to test the hypothesis that selective omission of axillary surgery in distinct responders after NACT will not deteriorate survival. In the planned trial, axillary surgery will be completely eliminated for initially cN0 TNBC and HER2-positive breast cancer patients who achieve pCR in breast after NACT determined by lumpectomy.

The trial is designed as a prospective, single-center, single-arm study with a limited number of patients (N=136). Patients will be recruited in China over a period of 36 months. Our results, together with other ongoing studies in other parts of the world with a similar design, might give practice-changing results and spare the time and the costs of a randomized comparison.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Core biopsy confirmed unicentric primary invasive triple-negative or HER2-positive breast cancer. Multifocal or multicentric tumors allowed only if breast-conserving surgery is deemed feasible.
* At least 18 years of age
* Initial tumor stage cT1c-T3N0M0 prior to NACT. cN0 stage established by clinical examination and ultrasonography
* In cases with suspicious lymph node, a negative core biopsy or fine needle aspiration (FNA) biopsy of the sonographically suspected lymph node is required
* Standard NACT with evident radiologic response
* Planned breast-conserving surgery with postoperative external whole-breast irradiation

Exclusion Criteria:

* History of previous malignancy
* Histologically proven N1 patients, patients with distant metastasis (M1)
* Pregnant or lactating patients
* Inflammatory breast cancer
* Radiologically non-responsive after NACT
* Mastectomy planned after NACT
* planned intraoperative radiotherapy (e.g. Intrabeam) or postoperative partial breast irradiation (e.g. multicatheter technique) alone; both procedures are allowed as boost techniques
* Written informed consent not obtained

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
ipsilateral axillary recurrence-free survival | 5-year
  time between randomization and confirmed ipsilateral axillary recurrence

SECONDARY OUTCOMES:
locoregional lymph node recurrence-free survival | 5-year
  time between randomization and confirmed locoregional lymph node recurrence
distant metastasis-free survival | 5-year
  time between randomization and confirmed distant metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China